CLINICAL TRIAL: NCT05463757
Title: Registration of Oral Hedgehog Inhibitors Vismodegib and Sonidegib in the Treatment of Advanced and Multiple Basal Cell Carcinoma in the Netherlands: a Prospective Registration Study.
Brief Title: Oral Hedgehog Inhibitors in the Treatment of Basal Cell Carcinoma in the Netherlands: a Prospective Registration Study
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: METC 2018-0452-A-10 Vismodegib
Record Dates: First submitted 2022-05-31; First posted 2022-07-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Basal Cell Carcinoma; Locally Advanced Basal Cell Carcinoma; Metastatic Basal Cell Carcinoma; Gorlin Syndrome; Basal Cell Nevus Syndrome; Carcinoma, Basal Cell; Carcinoma; Basal Cell Tumor; Skin Cancer; Neoplasm of Skin; Neoplasms, Basal Cell
Keywords: Oral hedgehog inhibitors; Vismodegib; Sonidegib; Erivedge; Odomzo
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome; Carcinoma; Neoplasms, Basal Cell; Skin Neoplasms | interventions — HhAntag691; sonidegib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Oral hedgehog inhibitor: Oral hedgehog inhibitors vismodegib (Erivedge) or sonidegib (Odomzo)
  Interventions: Drug: Vismodegib; Drug: Sonidegib

INTERVENTIONS:
Drug: Vismodegib — Oral vismodegib (Erivedge), taken daily or every other day (depending on doctor's description)
  Other Names: Erivedge
Drug: Sonidegib — Sonidegib (Odomzo), taken daily or every other day (depending on doctor's description)
  Other Names: Odomzo

SUMMARY:
Background: Oral hedgehog inhibitors vismodegib and sonidegib have been used for the treatment of locally advanced (laBCC), metastatic basal cell carcinoma (mBCC) and in basal cell nevus syndrome (BCNS) patients. In the Netherlands, targeted therapy with vismodegib and sonidegib has been available since 2013 and 2021, respectively. No direct comparative studies have been performed between the two oral hedgehog inhibitors (HHI) vismodegib and sonidegib yet . In addition, data for sonidegib are not yet available.

Objective: The aim of this study is 1) to evaluate the effectiveness of oral HHIs in the treatment of laBCC, mBCC and BCNS patients and 2) to compare the oral HHIs vismodegib and sonidegib.

Study design: prospective registration study that includes all patients, regardless of age and gender, with histologically proven basal cell carcinoma receiving treatment with either vismodegib or sonidegib in the Netherlands. Patient, tumor and treatment information was gathered from patient records.

Main study parameters/endpoints: The primary outcome for measuring efficacy/tumor response was median progression free survival (PFS) where the decrease, stagnation or increase in tumor size is measured by maximum diameter. Secondary outcomes are frequency, severity and reversibility of treatment-emergent adverse events and disease-specific quality of life expressed as mean scores on the EORTC-QLQ-C30 and aBCCdex questionnaires.

DETAILED DESCRIPTION:
This is a prospective registration study conducted in eight academic hospitals in the Netherlands. Vismodegib and sonidegib are currently only prescribed in academic hospitals in the Netherlands. Therefore, this multicenter approach with all academic centers in the Netherlands provides a complete insight into the prescription of these oral HHIs in the Netherlands. The study takes place at the dermatology and oncology department of Maastricht University Medical Center+ (MUMC+), Erasmus University Medical Center (Erasmus MC) Rotterdam, Netherlands Cancer Institute (NKI) Amsterdam, University Medical Center Groningen (UMCG), University Medical Center Utrecht (UMC Utrecht), Amsterdam University Medical Center (Amsterdam UMC), Radboud University Medical Center (Radboudumc) and Leiden University Medical Center (LUMC).

All patients receiving at least one dose of vismodegib or sonidegib for the treatment of basal cell carcinoma (laBCC, mBCC, multiple BCCs in BCNS and in non-BCNS) (in regular care) will be included, provided they give permission and sign the informed consent form. Treating physicians then systematically register data on treatment using a uniform registration format. This registration includes the effectiveness of the drug measured by tumor diameter*, adverse events according to the CTCAE version 5.0, and data such as age, gender, World health organization (WHO) status, scores on the G8 questionnaire, medication use, comorbidities, indication, dosage, treatment duration, laboratory values, and reason for discontinuation of treatment. In addition, twice a year scores on the EORTC-QLQ-C30 and aBCCdex questionnaires are registered. All data will be extracted from electronic patient files en will be entered anonymously in a Castor database.

The primary outcome for measuring efficacy/tumor response is median progression free survival (PFS) where the decrease, stagnation or increase in tumor size is measured by maximum tumor diameter*. Secondary outcomes are frequency, severity and reversibility of treatment-emergent adverse events and disease-specific quality of life expressed as mean scores on the EORTC-QLQ-C30 and aBCCdex questionnaires. In addition, the association of patient characteristics on drug efficacy and adverse events will be analysed.

*In case of gorlin goltz syndrome or multiple BCCs, at least 3 target lesions are registered whose diameters are monitored over time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* All ages
* Diagnosed with locally advanced basal cell carcinoma (laBCC), metastatic basal cell carcinoma (mBCC), multiple basal cell carcinomas or Gorlin syndrome
* Use of oral hedgehog inhibitor vismodegib or sonidegib

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All men and women, regardless of age, diagnosed with advanced basal cell carcinoma, metastatic basal cell carcinoma, multiple basal cell carcinomas or Gorlin syndrome, for which an oral hedgehog inhibitor (vismodegib or sonidegib) is used in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Median progression free survival | though study completion, an average of 3 years
  The main study outcome measure is the median progression free survival (PFS) where the decrease, stagnation or increase in tumor size is measured by maximum diameter.

SECONDARY OUTCOMES:
Adverse events | At baseline (start of treatment), after 1 month and every 3 months thereafter during use of vismodegib or sonidegib, at discontinuation of the treatment and 3 months after discontinuation of the treatment.
  Frequency, severity and reversibility of treatment-emergent adverse events, measured according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Disease-specific quality of life | At the start of treatment and every 6 months thereafter, until vismodegib or sonidegib is no longer used.
  Disease-specific quality of life expressed as mean scores on the validated European Organisation for Research and Treatment of Cancer (EORTC) core quality of life (EORTC-QLQ-C30) questionnaire.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Disease-specific quality of life | At the start of treatment and every 6 months thereafter, until vismodegib or sonidegib is no longer used.
  Disease-specific quality of life expressed as mean scores on the validated advanced basal cell carcinoma index (aBCCdex) questionnaire.
  The aBCCdex consists of 26 questions related to symptoms, emotions, worry, avoidance behavior and influence on daily life. Scales range in score from 1 to 7 and from 1 to 6. A higher score correlates with a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: K Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (8):
- Netherlands (8):
  - Radboudumc, Nijmegen, Gelderland
  - Maastricht University Medical Center +, Maastricht, Limburg
  - Amsterdam UMC, Amsterdam, North Holland
  - Netherlands Cancer Institute - AVL, Amsterdam, North Holland
  - UMCG, Groningen, Provincie Groningen
  - LUMC, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Verkouteren BJA, Wakkee M, Reyners AKL, Nelemans P, Aarts MJB, Racz E, Terra JB, Devriese LA, Alers RJ, Kapiteijn E, van Doorn R, Bekkenk MW, Reinders MGHC, Mosterd K. Eight years of experience with vismodegib for advanced and multiple basal cell carcinoma patients in the Netherlands: a retrospective cohort study. Br J Cancer. 2021 Mar;124(7):1199-1206. doi: 10.1038/s41416-020-01220-w. Epub 2021 Jan 19. PMID 33462360
- [Background] Sekulic A, Migden MR, Oro AE, Dirix L, Lewis KD, Hainsworth JD, Solomon JA, Yoo S, Arron ST, Friedlander PA, Marmur E, Rudin CM, Chang AL, Low JA, Mackey HM, Yauch RL, Graham RA, Reddy JC, Hauschild A. Efficacy and safety of vismodegib in advanced basal-cell carcinoma. N Engl J Med. 2012 Jun 7;366(23):2171-9. doi: 10.1056/NEJMoa1113713. PMID 22670903
- [Background] Basset-Seguin N, Hauschild A, Kunstfeld R, Grob J, Dreno B, Mortier L, Ascierto PA, Licitra L, Dutriaux C, Thomas L, Meyer N, Guillot B, Dummer R, Arenberger P, Fife K, Raimundo A, Dika E, Dimier N, Fittipaldo A, Xynos I, Hansson J. Vismodegib in patients with advanced basal cell carcinoma: Primary analysis of STEVIE, an international, open-label trial. Eur J Cancer. 2017 Nov;86:334-348. doi: 10.1016/j.ejca.2017.08.022. Epub 2017 Nov 5. PMID 29073584
- [Background] Dreno B, Kunstfeld R, Hauschild A, Fosko S, Zloty D, Labeille B, Grob JJ, Puig S, Gilberg F, Bergstrom D, Page DR, Rogers G, Schadendorf D. Two intermittent vismodegib dosing regimens in patients with multiple basal-cell carcinomas (MIKIE): a randomised, regimen-controlled, double-blind, phase 2 trial. Lancet Oncol. 2017 Mar;18(3):404-412. doi: 10.1016/S1470-2045(17)30072-4. Epub 2017 Feb 8. PMID 28188086
- [Background] Ben Ishai M, Tiosano A, Fenig E, Ben Simon G, Yassur I. Outcomes of Vismodegib for Periocular Locally Advanced Basal Cell Carcinoma From an Open-label Trial. JAMA Ophthalmol. 2020 Jul 1;138(7):749-755. doi: 10.1001/jamaophthalmol.2020.1539. PMID 32407451
- [Background] Dutch Society for Dermatology and Venereology (NVDV). Basal Cell Carcinoma: Dutch Guideline (Dutch Society for Dermatology and Venereology (NVDV). 2015).
- [Background] Xie P, Lefrancois P. Efficacy, safety, and comparison of sonic hedgehog inhibitors in basal cell carcinomas: A systematic review and meta-analysis. J Am Acad Dermatol. 2018 Dec;79(6):1089-1100.e17. doi: 10.1016/j.jaad.2018.07.004. Epub 2018 Jul 10. PMID 30003981
- [Background] Sekulic A, Migden MR, Basset-Seguin N, Garbe C, Gesierich A, Lao CD, Miller C, Mortier L, Murrell DF, Hamid O, Quevedo JF, Hou J, McKenna E, Dimier N, Williams S, Schadendorf D, Hauschild A; ERIVANCE BCC Investigators. Long-term safety and efficacy of vismodegib in patients with advanced basal cell carcinoma: final update of the pivotal ERIVANCE BCC study. BMC Cancer. 2017 May 16;17(1):332. doi: 10.1186/s12885-017-3286-5. PMID 28511673
- [Background] Sekulic A, Migden MR, Lewis K, Hainsworth JD, Solomon JA, Yoo S, Arron ST, Friedlander PA, Marmur E, Rudin CM, Chang AL, Dirix L, Hou J, Yue H, Hauschild A; ERIVANCE BCC investigators. Pivotal ERIVANCE basal cell carcinoma (BCC) study: 12-month update of efficacy and safety of vismodegib in advanced BCC. J Am Acad Dermatol. 2015 Jun;72(6):1021-6.e8. doi: 10.1016/j.jaad.2015.03.021. PMID 25981002
- [Background] Dummer R, Ascierto PA, Basset-Seguin N, Dreno B, Garbe C, Gutzmer R, Hauschild A, Krattinger R, Lear JT, Malvehy J, Schadendorf D, Grob JJ. Sonidegib and vismodegib in the treatment of patients with locally advanced basal cell carcinoma: a joint expert opinion. J Eur Acad Dermatol Venereol. 2020 Sep;34(9):1944-1956. doi: 10.1111/jdv.16230. Epub 2020 Mar 4. PMID 31990414
- [Background] Epstein EH. Basal cell carcinomas: attack of the hedgehog. Nat Rev Cancer. 2008 Oct;8(10):743-54. doi: 10.1038/nrc2503. PMID 18813320
- [Background] Lewis K, Dummer R, Farberg AS, Guminski A, Squittieri N, Migden M. Effects of Sonidegib Following Dose Reduction and Treatment Interruption in Patients with Advanced Basal Cell Carcinoma During 42-Month BOLT Trial. Dermatol Ther (Heidelb). 2021 Dec;11(6):2225-2234. doi: 10.1007/s13555-021-00619-4. Epub 2021 Oct 20. PMID 34669179
- [Background] Villani A, Costa C, Fabbrocini G, Ruggiero A, Scalvenzi M. Dose reduction during routine treatment of locally advanced basal cell carcinoma with the hedgehog inhibitor sonidegib to manage adverse effects: A retrospective case series. J Am Acad Dermatol. 2021 Apr;84(4):e211-e212. doi: 10.1016/j.jaad.2020.12.006. Epub 2020 Dec 7. No abstract available. PMID 33301802